CLINICAL TRIAL: NCT04045847
Title: A Clinical Study to Investigate the Safety, Tolerance and Efficacy Evaluation of Single-centre, Open-label of Local Treatment of CD147-CART in Recurrent Glioblastoma.
Brief Title: CD147-CART Cells in Patients With Recurrent Malignant Glioma.
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Chen Zhinan-2
Record Dates: First submitted 2019-08-04; First posted 2019-08-06 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2019-05

CONDITIONS: Recurrent Glioblastoma; CD147 Positive
Keywords: glioma; CD147; CAR-T
MeSH Terms: conditions — Glioblastoma; Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD147-CART (Experimental): CD147-CAR modified T cells, intracavity injection, 3+3 design with de-escalation in half step, every 7 days for 3 weeks
  Interventions: Biological: CD147-CART

INTERVENTIONS:
Biological: CD147-CART — Three doses of CD147-CART cells were injection to intracavity by Ommaya Reservoir.
  Other Names: anti-CD147 chimeric antigen receptor T cells

SUMMARY:
This is a single-center, single-arm, open label and dose escalation clinical study of anti-CD147 CART cells in patients with recurrent malignant glioma.

DETAILED DESCRIPTION:
Patients autologous T cells are activated and then engineered to express chimeric antigen receptors (CARs) specific for CD147(CD147-CART). CAR-T cells are expanded in culture and returned to the patient by Ommaya Reservoir at specific cell doses. Three CD147-CART doses patient are planned at 1-week intervals. Serum cytokine level and CAR-T cell number will be measured in whole treatment session.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 year and ≤ 65 years, both male and female;
2. Recurrent glioblastoma patients confirmed by histology or cytology, which have received standard care of STUPP protocol (TMZ concurrent chemoradiotherapy and adjuvant chemotherapy protocol) after surgery;
3. Cerebral ventricle was not opened after glioma surgery;
4. More than 6 months after the first glioma surgery;
5. Tumor lesions that can be evaluated or measured according to RANO criteria (Measurable enhancement lesions were defined as enhancement lesions with clear upper boundary of CT or MRI, capable of developing on ≥2 axial films with layer thickness of 5 mm, and the length and diameter of each other were >10 mm. If the scanning layer thickness is large, the minimum measurable lesion should be >2 times thick);
6. CD147+ was confirmed by histologically diagnosis (IHC staining).
7. Adequate PBMC can be obtained according to the requirements of cell preparation, and there are no other contraindications for lymphocyte collection;
8. KPS score ≥70;
9. Patient with a life expectancy of greater than three months;
10. Patients with entirely informed consent and voluntarily sign the informed consent by themselves or their legal representative.

Exclusion Criteria:

1. Patients who have received radiotherapy after recurrence;
2. Patients who have received corticosteroids or other immunosuppressive agents in the past 2 weeks;
3. Patients who have received live vaccine in the past 4 weeks and/or plan to receive live vaccine after participating in the trial;
4. Patients who have received chemotherapy in addition to lymphocyte clearance in the past 2 weeks;
5. Patients who have not recover from adverse events caused by previous anti-tumor therapy (≤1 according to CTCAE v5.0) prior to enrollment, except for hair loss；
6. Patients who have received gene therapy, cell therapy or immune therapy；
7. Patients who have received organ transplantation；
8. Patients who cannot able to perform craniocerebral MRI examination;
9. Patients with following abnormalities:

   1. Absolute neutrophil count (ANC)<1.5×109/L， platelet (PLT)<80×109/L or hemoglobin(HGB)<100 g/dL；
   2. Prothrombin time (PT), activated partial thromboplastin time (APTT) or international normalized ratio (INR) > 1.5×ULN (upper normal value);
   3. Total bilirubin(TBIL) > 2×ULN; ALT, AST or ALP>3×ULN;
   4. Serum creatinine (Cr)≥1.5×ULN or glomerular filtration rate (GFR) < 60mL/min×1.73m2；
   5. Syphilis test (TRUST) positive, Anti-HIV positive, Anti-HCV positive with HCV-RNA level higher than the lower limit of detection (LOD), or HBcAb positive with HBV-DNA level higher than the LOD;
   6. Left ventricular ejection fraction (LVEF) < 50%;
10. An acute bacterial or fungal infection that requires intravenous antibiotics during CAR-T cell therapy;
11. Patients who presented with negligent compensatory heart failure (NYHA grade III and IV), unstable angina pectoris, acute myocardial infarction, persistent and clinically significant arrhythmia within 3 months;
12. Patients who requires supplemental oxygen to keep saturation greater than 95% and the situation is not expected to resolve within 2 weeks;
13. Patients with other malignant tumors that have not been effectively controlled within the past five years;
14. Patients who suffering from tuberculosis and not cured;
15. Patients with a history of allergic reactions attributed to any agents or compounds involved in this study;
16. Patients allergic to contrast agents;
17. Patients with a history of mental disorders;
18. Patients with a history of drug abuse;
19. Pregnant and lactating women, or planning to become pregnant during the study;
20. Patients of childbearing age who unwilling or unable to use effective and adequate contraception during and 3 months after the study;
21. Patients who enrolled in other clinical trials within 30 days;
22. Patients who were considered not suitable for this clinical trial by investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2019-05-30 (Actual); Primary Completion 2020-10-30 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and type of adverse events induced by CD147-CART | 12 weeks
  To assess the safety and tolerability of CD147-CART (anti-CD147 CAR-T cell) for glioma which measured by number and type of adverse events.

SECONDARY OUTCOMES:
DLT and MTD of CD147-CART cell | 12 weeks
  To determine the dose limited toxicity (DLT) and maximum tolerated dose (MTD) of CD147-CART.
Clinical Activity of CD147-CART cell | 2 years
  To evaluate treatment response of CD147-CART for glioma
CD147-CART detection in Peripheral Blood | 2 years
  Quantification of CD147-CART cells in blood samples.

CONTACTS AND LOCATIONS:
Locations (1):
- National Translational Science Center for Molecular Medicine & Department of Cell Biology, Xi'an, Shaanxi, China